CLINICAL TRIAL: NCT02340195
Title: Interventional, Single-site, Open-label, Reduced/Staged, Multiple-dose Study Investigating the Pharmacokinetic Properties of Idalopirdine (Lu AE58054) in Patients With Renal Impairment and in Healthy Subjects
Brief Title: Pharmacokinetic Properties of Idalopirdine (Lu AE58054) in Subjects With and Without Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14916A; 2012-005647-25 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer Disease
Keywords: Kidney impairment
MeSH Terms: conditions — Alzheimer Disease; Renal Insufficiency | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Idalopirdine (Lu AE58054) 60 mg (Group A) (Experimental): 8 patients with severe renal impairment and not on dialysis
  Interventions: Drug: Idalopirdine (Lu AE58054) 60 mg
- Idalopirdine (Lu AE58054) 60 mg (Group B) (Experimental): 8 healthy subjects
  Interventions: Drug: Idalopirdine (Lu AE58054) 60 mg
- Idalopirdine (Lu AE58054) 60 mg (Group C) (Experimental): Group C will not be tested, if severe renal impairment does not alter the pharmacokinetics to a clinically relevant extent, based on results from group A and B
  8 patients with moderate renal impairment
  Interventions: Drug: Idalopirdine (Lu AE58054) 60 mg
- Idalopirdine (Lu AE58054) 60 mg (Group D) (Experimental): Group D will not be tested, if severe renal impairment does not alter the pharmacokinetics to a clinically relevant extent, based on results from group A and B
  8 patients with mild renal impairment
  Interventions: Drug: Idalopirdine (Lu AE58054) 60 mg

INTERVENTIONS:
Drug: Idalopirdine (Lu AE58054) 60 mg — encapsulated film-coated tablets for oral use once daily for 10 days

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics properties of idalopirdine following multiple dosing in patients with renal impairment and compare to those in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 50 and 75 years (inclusive)
* BMI ≥18.5 kg/m2 and ≤32 kg/m2 at the Screening Visit.
* Group A: Patients with severe renal impairment renal impairment (creatinine clearance (ClCr) ≤29 mL/min)
* Group B: Healthy subjects with normal kidney function (creatinine clearance (ClCr) ≥90 mL/min, inclusive)
* Group C: Patients with moderate renal impairment ((creatinine clearance between 30 - 59 mL/min, inclusive)
* Group D: Patients with mild renal impairment (Creatinine clearance between 60 - 89 mL/min, inclusive)

Exclusion Criteria:

•The subject has taken disallowed medication <1 week prior to the first dose of IMP or <5 half-lives prior to the first dose of IMP for any disallowed medication taken, whichever is longer)

Other protocol defined inclusion and exclusion criteria do apply

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Area under the LuAE58054 plasma concentration-time curve from time zero to 24h(AUC0-24) | Day 10
Maximum observed concentration (Cmax) of Lu AE58054 | 0-12 hours day 10

CONTACTS AND LOCATIONS:
Locations (1):
- DE801, München, Germany